CLINICAL TRIAL: NCT01505361
Title: Oral Administration of a Probiotic Strain to Pregnant Women: Effects on the Prevention of Lactational Mastitis and on the Eradication of GBS Colonization
Brief Title: Study of a Probiotic Strain to Prevent Mastitis and to Eradicate GBS Colonization
Acronym: PROBIOPREG
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Juan M. Rodríguez, Professor, PhD, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PROBIOPREG
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Mastitis
Keywords: probiotic; Lactobacillus salivarius; mastitis; prevention; group B streptococci; intrapartum prophylaxis
MeSH Terms: conditions — Mastitis | interventions — Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Pregnant women at 30 week of pregnancy(n=50) receiving Lactobacillus salivarius PS2(9 log per day, until birth)
  Interventions: Biological: Lactobacillus salivarius PS2
- Placebo (Placebo Comparator): Pregnant women at 30 week of pregnancy(n=50) receiving the excipient (once a day, until birth)
  Interventions: Biological: Excipient (milk powder)

INTERVENTIONS:
Biological: Lactobacillus salivarius PS2 — 9 log10 (colony-forming units), freeze-dried powder, daily for 30 week of pregnancy until birth
  Arms: Probiotic
Biological: Excipient (milk powder) — 100 mg/once a day from 30 week of pregnancy until birth
  Arms: Placebo

SUMMARY:
In previous studies, the investigators have seen that carefully-selected Lactobacillus strains are a good alternative to antibiotics for the treatment of lactational mastitis. The objective of this new study is to check if they can also have a preventive role when administered to women with a history of mastitis with one or more previous infants. Since the investigators have also realized that peripartum antibiotherapy (mainly GBS-targeting intrapartum prophylaxis)is a predisposing factor for mastitis (because of the selection of resistant bacteria), the investigators would also like to test if administration of the strains to GBS-colonized pregnant women may lead to GBS eradication. Therefore, a mastitis-predisposing factor would de avoid.

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnancy
* Healthy women
* Lactational mastitis in, at least, a previous lactation period
* No symptomatic vaginal infections

Exclusion Criteria:

* Any kind of health problems related to pregnancy
* Symptomatic vaginal infections
* Allergy to cow's milk protein
* Intolerance to lactose
* Antibiotic treatment

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinical mastitis confirmed by microbiological cultures and somatic cell counts | Weekly during the first 6 months after birth

SECONDARY OUTCOMES:
Evidence of eradication og GBS colonization as confirmed by microbiological analysis of vaginal exudate and rectal swab | At weeks 30, 35, 40 of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Rodriguez, PhD, Principal Investigator — Complutense University of Madrid, Spain
Locations (1):
- Public Primary Health Care Centers network, Madrid, Madrid, Spain

REFERENCES:
- [Background] Arroyo R, Martin V, Maldonado A, Jimenez E, Fernandez L, Rodriguez JM. Treatment of infectious mastitis during lactation: antibiotics versus oral administration of Lactobacilli isolated from breast milk. Clin Infect Dis. 2010 Jun 15;50(12):1551-8. doi: 10.1086/652763. PMID 20455694
- [Background] Jimenez E, Fernandez L, Maldonado A, Martin R, Olivares M, Xaus J, Rodriguez JM. Oral administration of Lactobacillus strains isolated from breast milk as an alternative for the treatment of infectious mastitis during lactation. Appl Environ Microbiol. 2008 Aug;74(15):4650-5. doi: 10.1128/AEM.02599-07. Epub 2008 Jun 6. PMID 18539795
- [Derived] Crepinsek MA, Taylor EA, Michener K, Stewart F. Interventions for preventing mastitis after childbirth. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD007239. doi: 10.1002/14651858.CD007239.pub4. PMID 32987448
- [Derived] Fernandez L, Cardenas N, Arroyo R, Manzano S, Jimenez E, Martin V, Rodriguez JM. Prevention of Infectious Mastitis by Oral Administration of Lactobacillus salivarius PS2 During Late Pregnancy. Clin Infect Dis. 2016 Mar 1;62(5):568-573. doi: 10.1093/cid/civ974. Epub 2015 Nov 26. PMID 26611780